CLINICAL TRIAL: NCT02975687
Title: CD19 CAR T Cells in Patients With Resistant or Refractory CD19+ Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Juventas Cell Therapy Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QT2016002; HY001001 (Other: Juventas Cell Therapy Ltd.)
Record Dates: First submitted 2016-11-23; First posted 2016-11-29 (Estimated); Last update posted 2025-06-03 (Actual); Status verified 2019-07

CONDITIONS: Acute Lymphoblastic Leukemia, Adult B-Cell; Acute Lymphoblastic Leukaemia Recurrent
Keywords: Acute; Leukemia; Lymphoid; CD19; Refractory
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia

ARMS (1):
- Arm A (Experimental): CD19 CAR T cells will be administered by i.v. injection as a using a "split dose" (total dose of 5x10^6/kg-5x10^7/kg) approach to dosing:10% on day 0, 30% on day 1 and 60% on day 2.
  Interventions: Biological: CD19 CAR T cells

INTERVENTIONS:
Biological: CD19 CAR T cells — CD19 CAR T cells was transduced with a lentiviral vector to express anti-CD19 scFv TCRζ:4-1BB.

SUMMARY:
In this single-center, open-label, no control, prospective clinical trial, a total of 20 resistant or refractory CD19+ B cell acute lymphoblastic leukemia (ALL) patients will be enrolled. CD19 CAR T cells will be administered by i.v. injection as a using a "split dose" (total dose of 5x10^6/kg-5x10^7/kg) approach to dosing:10% on day 0, 30% on day 1 and 60% on day 2. The purpose of current study is to determine the clinical efficacy and safety of CD19 CAR T cells in patients with chemotherapy resistant or refractory CD19+ ALL.

DETAILED DESCRIPTION:
In this single-center, open-label, nonrandomized, no control, prospective clinical trial, a total of 20 resistant or refractory CD19+ B cell acute lymphoblastic leukemia (ALL) patients will be enrolled. Patients will be diagnosed according to morphologic, immunologic, cytogenetic and molecular(MICM) criteria, including bone marrow morphology, immunophenotype, cytogenetic and molecular examination. CD19 CAR T cells transduced with a lentiviral vector to express anti-CD19 scFv TCRζ:4-1BB,administered by i.v. injection as a using a "split dose" (total dose of 5x10^6/kg-5x10^7/kg) approach to dosing:10% on day 0, 30% on day 1 and 60% on day 2. This protocol will be given to subjects with unmet medical needs for which there are no effective therapies known at this time. Side effects of CD19 CAR T cells therapy will be monitored. The purpose of current study is to determine the clinical efficacy and safety of CD19 CAR T cells therapy in patients with chemotherapy resistant or refractory CD19+ ALL.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 70 years with relapsed or refractory CD19 positive ALL(ie, ≥20% blasts CD19-positive) due to receive either salvage 1 or salvage 2 therapy. Ph+ ALL patients must have failed treatment with at least 1 second generation tyrosine kinase inhibitor.
* Bone marrow involvement with≥20% lymphoblasts.
* Eastern Cooperative Oncology Group (ECOG) Performance status 0-2.
* Adequate end organ function as defined by: Total bilirubin ≤ 1.5 x upper limit of normal（ULN）; serum glutamic-oxaloacetic transaminase(SGOT) and serum glutamic pyruvic transaminase(SGPT) ≤ 2.5 x ULN; Creatinine ≤ 1.5 x ULN or any serum creatinine level associated with a measured or calculated creatinine clearance of ≥ 40ml/min.
* Patients should sign informed consent form.

Exclusion Criteria:

* Isolated extramedullary relapse.
* Active central nervous system leukemia.
* Prior chemotherapy within ≤2 weeks before enrollment with the following exceptions: steroids, hydroxyurea, oral mercaptopurine, methotrexate, vincristine, thioguanine, and tyrosine kinase inhibitors are permitted within 2 weeks of enrollment as maintenance or to reduce the peripheral blood blast count. Patients must have recovered from acute toxicity of all previous therapy prior to enrollment.
* Prior allogeneic hematopoietic stem cell transplant (HSCT) ≤ 4 months before enrollment. Patients must have completed immunosuppression therapy prior to enrollment. At enrollment, patients must not have > grade 2 acute GVHD, or either moderate or severe limited chronic GVHD, or extensive GVHD of any severity.
* Peripheral lymphoblasts > 10,000/μl (treatment with hydroxyurea and/or steroids is permitted within 2 weeks of enrollment to reduce the WBC count).
* Known systemic vasculitides, primary or secondary immunodeficiency(such as HIV infection or severe inflammatory disease).
* Major surgery within ≤ 4 weeks before enrollment.
* Impaired cardiac function:Ejection fraction < 45 % on MUGA scan. QTc interval > 450 msec on baseline ECG (using the QTcB formula). If QTcB interval>450 msec and electrolytes are not within normal ranges, electrolytes should be corrected and then the patient re-screened for QTc. Myocardial infarction within 6 months prior to starting study; other clinically significant heart disease (e.g. unstable angina, congestive heart failure or uncontrolled hypertension, uncontrolled arrhythmias).
* Administration of live vaccine ≤ 4 weeks before enrollment.
* Other concurrent severe and/or uncontrolled medical conditions:

Patients with another primary malignant disease, except those that do not currently require treatment; acute or chronic liver, pancreatic or severe renal disease; another severe and/or life-threatening medical disease.

* Evidence of uncontrolled current serious active infection.
* Patients who are: (a) pregnant, (b) breast feeding, (c) of childbearing potential without a negative pregnancy test prior to baseline and (d) male or female of childbearing potential unwilling to use contraceptive precautions throughout the trial (post-menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential).
* Who is known human deficiency virus (HIV) positive.
* Use of any other investigational agent in the last 30 days.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-11; Primary Completion 2018-12 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
The complete remission (CR) rate | Participants will be followed for the duration of the treatment, an expected average of 12 months.

SECONDARY OUTCOMES:
Disease-free survival (DFS) | From the date of complete remission(CR) until the date of documented relapse,assessed up to 60 months.
Number of adverse event of CD19 CAR T cells treatment | Participants will be followed for the duration of the treatment, an expected average of 24 months.
Grade of adverse event of CD19 CAR T cells treatment | Participants will be followed for the duration of the treatment, an expected average of 24 months.
Duration of in vivo survival of CD19 CAR T cells. | Participants will be followed for the duration of the treatment, an expected average of 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jianxiang Wang, Dr., Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, China

REFERENCES:
- [Derived] Gu R, Liu F, Zou D, Xu Y, Lu Y, Liu B, Liu W, Chen X, Liu K, Guo Y, Gong X, Lv R, Chen X, Zhou C, Zhong M, Wang H, Wei H, Mi Y, Qiu L, Lv L, Wang M, Wang Y, Zhu X, Wang J. Efficacy and safety of CD19 CAR T constructed with a new anti-CD19 chimeric antigen receptor in relapsed or refractory acute lymphoblastic leukemia. J Hematol Oncol. 2020 Sep 7;13(1):122. doi: 10.1186/s13045-020-00953-8. PMID 32894185